CLINICAL TRIAL: NCT05500703
Title: Brain Regions and Functional Neuronal Network Characteristics of Dexmedetomidine Analgesia Under Intraoperative fMRI
Brief Title: Brain Regions and Functional Neuronal Network Characteristics of Dexmedetomidine Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CINI-AD-20220706
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy; Radiofrequency Ablation; Intracranial Surgery
MeSH Terms: conditions — Epilepsy | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): 1.5 µg kg-1 h-1 dexmedetomidine
  Interventions: Drug: Dexmedetomidine Injectable Solution
- Placebo group (Placebo Comparator): 0.9% sodium chloride injection
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Solution — continuous pump of 1.5ug / kg / h Dexmedetomidine 15min before anesthesia induction, continuous infusion for 30min after anesthesia induction, and then nuclear magnetic scanning was started.
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine group
Drug: Sodium Chloride 0.9% Inj — the equivalent Sodium Chloride 0.9% Inj was continuously pumped before anesthesia induction, induced by opioids for 15min, and intraoperative fMRI scanning was started after continuous infusion for 30min.
  Other Names: only opioid and Sodium Chloride as placebo administration
  Arms: Placebo group

SUMMARY:
Background: Dexmedetomidine (Dex) is a highly selective 2-adrenergic receptor agonist with significant analgesia affection. This study is planned to explore the brain regions and functional neuronal network involved in promoting analgesia of Dexmedetomidine. Methods: Select 28 patients with the proposed intraoperative MR-guided radiofrequency ablation of epilepsy. The subjects were randomized into the Dexmedetomidine group (Dex group) (n=14) and the Placebo group (PO group) (n=14). DEX group: continuous intravenously administered 1.5 µg kg-1 h-1 dexmedetomidine 15min before anesthesia induction, continuous infusion for 15min after anesthesia induction, and then Intraoperative functional magnetic resonance imaging scanning was started. PO group: the equivalent administered speed 0.9% sodium chloride was continuously pumped for 15min before anesthesia induction, then induce and intraoperative fMRI scanning started after continuous 30min infusion. The intraoperative fMIR scan results were compared and analyzed to find the unique analgesic brain regions of DEX, and the differences of the functional neuronal network of analgesia effect between the two groups.

DETAILED DESCRIPTION:
Background: Dexmedetomidine (DEX) is a highly selective 2-adrenergic receptor agonist with significant analgesia affection. This study is planned to explore the brain regions and functional neuronal network involved in promoting analgesia of Dexmedetomidine. Methods: Select 12 patients with the proposed intraoperative MR-guided radiofrequency ablation of epilepsy. The subjects were randomized into the Dexmedetomidine group (DEX group) (n=14) and the Placebo group (PO group) (n=14). DEX group: continuous intravenously administered 1.5 µg kg-1 h-1 dexmedetomidine 15min before anesthesia induction, continuous infusion for 15min after anesthesia induction, and then Intraoperative functional magnetic resonance imaging scanning was started. OPI group: the equivalent administered speed 0.9% sodium chloride was continuously pumped for 15min before anesthesia induction, then induce and intraoperative fMRI scanning started after continuous 30min infusion. The intraoperative fMIR scan results were compared and analyzed to find the unique analgesic brain regions of DEX, and the differences of the functional neuronal network of analgesia effect between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of epilepsy and eligible for radiofrequency ablation
2. 20-50 years old;
3. American Society of Anesthesiologists rated (ASA) I-II
4. body mass index (BMI)18.5~27.9 kg·m2.

Exclusion Criteria:

1. pre-existing neuropsychiatric disorders;
2. emergency surgery;
3. coma;
4. depression;
5. cognitive impairment;
6. implanted with metal devices.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Measurement of analgesia relative brain regions assessed by BOLD under fMRI scanning | during operation
  Measurement of analgesia relative brain regions inDexmedetomidine group (DEX group) and the Opioid group (OPI group) assessed by BOLD under fMRI scanning, and compare the two group different at the same time

SECONDARY OUTCOMES:
Measurement of analgesia relative brain regions assessed by T1-MPRAGE under fMRI scanning | during operation
  Measurement of analgesia relative brain regions inDexmedetomidine group (DEX group) and the Opioid group (OPI group) assessed by T1-MPRAGE under fMRI scanning, and compare the two group different at the same time
Measurement of analgesia relative brain regions assessed by T2-SPACE under fMRI scanning | during operation
  Measurement of analgesia relative brain regions inDexmedetomidine group (DEX group) and the Opioid group (OPI group) assessed by T2-SPACE under fMRI scanning, and compare the two group different at the same time
systolic blood pressure (SBP) | during operation
  hemodynamic change of the two groups included systolic blood pressure (SBP)
diastolic blood pressure (DBP) | during operation
  hemodynamic change of the two groups included diastolic blood pressure (DBP)
mean arterial pressure (MAP) | during operation
  hemodynamic change of the two groups included mean arterial pressure (MAP)
heart rate (HR) | during operation
  hemodynamic change of the two groups included heart rate (HR)
NRS | Hour 4, Hour 12, Hour48 post-operatively
  NRS immediately after operation at rest.(The p-NRS was an 11-point scale with 0 indicating no pain and 10 equaled worst possible pain)

OTHER OUTCOMES:
PONV | Day 7 postoperatively
  modified postoperative nausea vomiting (PONV) score

CONTACTS AND LOCATIONS:
Overall Officials: Xinya Wang, Dr, Study Chair — China International Neuroscience Institute
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No